CLINICAL TRIAL: NCT04050345
Title: Tracking Mutations in Cell Free Tumour DNA to Predict Relapse in Early Colorectal Cancer
Acronym: TRACC
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4344
Record Dates: First submitted 2018-10-30; First posted 2019-08-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE tumour tissue will be retrieved from surgery of patients with stage I, II and III CRC and targeted resequencing by a clinically validated method for a panel of pre-specified genes such as KRAS, NRAS, BRAF, PIK3CA, TP53 and APC will be performed. The study will also collect plasma from these patients and extract cfDNA. ddPCR assays will be used to detect and track tumour specific mutations in cfDNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Part B TRACC Colon: Patients with diagnosis of large bowel cancer (in the colon) and no evidence of metastatic disease
- Part B TRACC Rectal: Patients who have a diagnosis of large bowel cancer (in the Rectum) and no evidence of metastatic disease
- Part C TRACC- Standard of Care Adjuvant Chemotherapy: Randomised to Arm A: Standard of Care Arm (Patients with fully resected high risk stage II or stage III colon or Rectal cancer with no evidence of metastatic disease. Patients with locally advanced rectal cancer who have previously undergone chemoradiotherapy are also eligible to enrol.
- Part C-ct DNA Guided Arm: Patients with fully resected high risk stage II or stage III colon or rectal cancer with no evidence of metastatic disease. Patients with locally advanced rectal cancer who have previously undergone chemoradiotherapy are also eligible to enrol.
  De-escalation of adjuvant chemotherapy in patients who have a post-operative ctDNA negative result

SUMMARY:
TRACC Part B This is a multi-centre, prospective, translational research study involving the collection and analysis of tumour tissue, serial blood samples and clinical data in patients with newly diagnosed stage I, II and III CRC.

TRACC Part C is a : (multi-centre, prospective, randomised study, of ctDNA guided adjuvant chemotherapy versus standard of care adjuvant chemotherapy study after curative surgery in patients with high risk stage II or stage III CRC. )It aims to demonstrate that a de-escalation strategy of ctDNA guided adjuvant chemotherapy is non- inferior to standard of care treatment as measured by 3 year disease free survival (DFS) in patients with high risk stage II or stage III colorectal cancer CRC with no evidence of minimal residual disease (MRD) (ctDNA negative)

DETAILED DESCRIPTION:
TRACC Part B: Despite potentially curative surgery +/- adjuvant chemotherapy, a proportional of patients with early stage CRC will experience disease relapse. Current tools for surveillance, e.g., blood sampling for tumour markers (CEA) are neither sensitive nor specific. We hypothesise that detection of mutations in circulating free DNA (cfDNA) in plasma can predict relapse in patients with early stage CRC.

Circulating cell free tumour DNA (ctDNA) maintains the same mutations that are present in tumour. In colorectal cancer CRC, primary tumours and& metastases exhibit high genomic concordance. Therefore the TRACC study TRACC Part B is investigating whether serial blood samples taken from in patients with stage II and III fully resected early stage CRC colorectal cancer that have undergone potentially curative surgery, blood samples to can be used to detect and& quantify ctDNA may in order to identify minimal residual disease MRD and predict relapse earlier than existing methods. CtDNA may ultimately help identify a subset of patients that are or are unlikely to benefit from adjuvant chemotherapy and could therefore safely spare some patients from receiving unnecessary chemotherapy & its associated side-effects.

TRACC Part C: We hypothesis that ctDNA guided adjuvant chemotherapy administration will enable biomarker driven selection of patients who would and would not benefit from adjuvant chemotherapy and thereby reduce the proportion of patient receiving unnecessary adjuvant chemotherapy, reducing the potential side effects associated with it, but without compromising disease free survival (DFS). : This part of the study will use tThe blood test ctDNA result from a post-operative blood sample willto guide adjuvant chemotherapy treatment decisions. The study aims to demonstrate that athe de -escalation strategy of ctDNA guided adjuvant chemotherapy is non-inferior to standard of care treatment as measured by 3 year DFS in patients with high risk stage II and stage III CRC, in those who have no evidence of MRD (ctDNA negative). after surgery for patients with colorectal cancer who are following the standard of care pathway. Patients are randomised at the post- operative time point to: Arm A (standard of care adjuvant chemotherapy), or Arm B (ctDNA guided adjuvant chemotherapy) arm. For the ct DNA guided arm, patients who are ctDNA negative at this time point will have their chemotherapy de-escalated.

ELIGIBILITY:
TRACC Part B Inclusion Criteria:

* New diagnosis of histologically confirmed CRC scheduled to undergo surgery with curative intent, with no radiological evidence of metastatic disease.
* Patients with high grade dysplasia whose imaging is suggestive of colorectal carcinoma (CRC) will be included but will be excluded post-surgery if carcinoma diagnosis is not confirmed
* Age≥18
* Ability to give informed consent
* Able to adhere to follow up schedule

TRACC Part B Exclusion Criteria:

* Scheduled to have neoadjuvant chemotherapy, (neoadjuvant chemoradiotherapy for patients with rectal cancer is permitted)
* Current or previous other malignancy within 5 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix or other non-invasive malignancy

TRACC Part C

Inclusion Criteria:

1. Subject ≥ 18 years of age
2. Subjects with histologically proven high risk stage II or stage III colon or rectal cancer treated with curative intent with surgery alone (any T, N1 or N2) with no evidence of metastatic disease. High risk stage II is defined as having one or more of the following: T4 disease, obstruction and/or perforation of the primary tumour during the pre-operative period, inadequate nodal harvest as indicated by <12 nodes examined, poorly differentiated grade on histology, perineural invasion, peritoneal involvement or extramural venous/lymphatic invasion. Subjects must be due to receive adjuvant chemotherapy after surgery or Subjects with histologically proven locally advanced stage III rectal cancer treated with neoadjuvant chemoradiotherapy (any T, N1 or N2, M0) with no evidence of metastatic disease are eligible. Subjects must be due to receive adjuvant chemotherapy after surgery
3. Fully surgically resected tumour with clear resection margins (i.e., >1 mm).
4. Adequate organ function

   * Absolute neutrophil function ≥1.0 x 109/ L
   * Platelet Count ≥ 75 x 109 / L
   * Haemoglobin ≥80g/L (blood transfusion before randomisation is allowed)
   * Adequate renal function (GFR ≥ 50ml/min if single agent capecitabine or CAPOX being administered) as calculated by Cockcroft and Gault equation
   * Aspartate aminotransferase/ Alanine aminotransferase levels ≤ 2.5 upper limit of normal
5. Absence of major post-operative complications or other clinical conditions that, in the opinion of the investigator, would contraindicate adjuvant chemotherapy
6. Patients should be assessed by Oncology team for suitability and assessment for adjuvant chemotherapy, be able to have post-operative ctDNA sample collected and be randomised by week 8 ± 2 weeks after surgery.
7. ECOG performance status 0- 2
8. Able to give informed consent

TRACC Part C Exclusion criteria

1. History of concurrent and previous malignancy within the last 5 years, with the exception of non- melanomatous skin cancer and carcinoma in situ 2. Any major post-operative complications or other clinical conditions that in the opinion of the investigator would contra-indicate adjuvant chemotherapy 3. Any subject not due to receive adjuvant chemotherapy will not be eligible for Part C of the study 4. Hypersensitivity or contraindication to the drug(s) associated with the planned choice of systemic chemotherapy (CAPOX or single agent capecitabine) as stated in the SmPC for each of the drugs 5. Subjects due to receive 5-Flurouracil (5-FU) based adjuvant chemotherapy (either single agent 5-FU or in combination with oxaliplatin) will not be eligible for Part C of the study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TRACC Part B patients will have eligibility assessed, prior to surgery and again post-operatively with the histopathology report from surgery using the criteria below. Patients meeting the eligibility criteria at the first assessment will be registered. Rectal cancer patients that undergo pre-operative radiotherapy or chemo-radiotherapy have an additional eligibility assessment after treatment with the results of their imaging.
  TRACC Part C: patients with histologically proven High risk Stage 2 or Stage 3 colon or rectal cancer, treated with curative surgery with no evidence of metastatic disease. Patients with histologically proven rectal cancer who have previously undergone neoadjuvant chemoradiotherapy are also eligible. Patients must be due to receive adjuvant chemotherapy,
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12-05 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
TRACC Part B (Translational sub study) | 6 years
  • To assess whether detection of ctDNA predicts for relapse in patients with stage II and III colorectal cancer (CRC) that have undergone surgery with curative intent
TRACC Part C (Randomised ctDNA guided adjuvant chemotherapy versus SoC study): | 4 years
  • To demonstrate de-escalation strategy of ctDNA guided adjuvant chemotherapy is non- inferior to standard of care treatment as measured by 3 year disease free survival in patients with high risk stage II or stage III colorectal cancer with no evidence of minimal residual disease (ctDNA negative)

SECONDARY OUTCOMES:
Relationship between ctDNA detection before, during and after treatment | 8 years
  To calculate the association between detectable ctDNA with disease free survival and overall survival at four time points during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Study Chair — Royal Marsden NHS Foundation Trust
Locations (71):
- United Kingdom (71):
  - Milton Keynes General Hospital, Milton Keynes, Buckinghamshire
  - Croydon University Hospital, Thornton Heath, Croydon
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset
  - Poole Hospital, Poole, Dorset
  - Broomfield Hospital, Chelmsford, Essex
  - Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - University Hospital of South Manchester & Manchester Royal Infirmary, Wythenshawe, Manchester
  - Musgrove Park Hospital, Taunton, Somerset
  - Weston General Hospital, Weston-super-Mare, Somerset
  - Epsom and St Helier's Hospitals NHS Trust, Carshalton, Surrey
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Guy's & St Thomas Hospital, London, UK
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Salisbury District Hospital, Salisbury, Whiltshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Bronglais Hospital, Aberystwyth
  - Stoke Mandeville Hospital, Aylesbury
  - Basildon and Thurrock University Hospitals, Basildon
  - Basingstoke and North Hampshire Hospitals, Basingstoke
  - Bedford Hospital, Bedford
  - Royal Blackburn Teaching Hospital, Blackburn
  - Pilgrim Hospital, Boston
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Burnley General Teaching Hospital, Burnley
  - West Suffolk Hospital, Bury
  - Addenbrookes Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - North Cumbria University Hospitals, Carlisle
  - Glangwili Hospital, Carmarthen
  - Castle Hill Hospital, Cottingham
  - University Hospitals Coventry & Warwickshire, Coventry
  - Leighton Hospital, Crewe
  - University Hospital Crosshouse, Crosshouse
  - Medway NHS Foundation Trust, Gillingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Princess Alexandra Hospital NHS Trust, Harlow
  - Withybush General Hospital, Haverfordwest
  - Wycombe Hospital, High Wycombe
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - Airedale General Hospital, Keighley
  - Kettering General Hospital, Kettering
  - Kingston Hospital Foundation Trust, Kingston upon Thames
  - Forth Valley Royal Hospital, Larbert
  - St James's University Hospital, Leeds
  - Lincoln County Hospital, Lincoln
  - Prince Philip Hospital, Llanelli
  - Barts Health NHS Trust, London
  - North Middlesex University Hospital NHS Trust, London
  - Royal Free Hospital, London
  - St George's NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust - London, London
  - Chelsea and Westminster, London
  - Maidstone & Tunbridge Wells NHS Trust, Maidstone
  - Chase Farm Hospital, Middlesex
  - Northampton General Hospital NHS Trust, Northampton
  - Nottingham University Hospital, Nottingham
  - George Eliot Hospital, Nuneaton
  - Royal Preston Hospital, Lancashire Teaching Hospitals, Preston
  - Barking Havering and Redbridge NHS Foundation Trust (Queen's Hospital, Romford
  - Weston Park Hospital, Sheffield
  - Royal Shrewsbury Hospital, Shrewsbury
  - South Tyneside District Hospital, South Shields
  - University Hospital Southampton, Southampton
  - Stockport NHS Foundation Trust, Stockport
  - Sunderland Royal Hospital, Sunderland
  - King's Mill Hospital, Sutton in Ashfield
  - Singleton Hospital, Swansea
  - Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan
  - Royal Hampshire County Hospital, Winchester

REFERENCES:
- [Derived] Slater S, Bryant A, Aresu M, Begum R, Chen HC, Peckitt C, Lazaro-Alcausi R, Carter P, Anandappa G, Khakoo S, Melcher L, Potter V, Marti FM, Huang J, Branagan G, George N, Abulafi M, Duff S, Raja A, Gupta A, West N, Bucheit L, Rich T, Chau I, Cunningham D, Starling N; TRACC Part B trial investigators. Tissue-Free Liquid Biopsies Combining Genomic and Methylation Signals for Minimal Residual Disease Detection in Patients with Early Colorectal Cancer from the UK TRACC Part B Study. Clin Cancer Res. 2024 Aug 15;30(16):3459-3469. doi: 10.1158/1078-0432.CCR-24-0226. PMID 38864835
- [Derived] Slater S, Bryant A, Chen HC, Begum R, Rana I, Aresu M, Peckitt C, Zhitkov O, Lazaro-Alcausi R, Borja V, Powell R, Lowery D, Hubank M, Rich T, Anandappa G, Chau I, Starling N, Cunningham D. ctDNA guided adjuvant chemotherapy versus standard of care adjuvant chemotherapy after curative surgery in patients with high risk stage II or stage III colorectal cancer: a multi-centre, prospective, randomised control trial (TRACC Part C). BMC Cancer. 2023 Mar 20;23(1):257. doi: 10.1186/s12885-023-10699-4. PMID 36941575